CLINICAL TRIAL: NCT06464172
Title: The GABAergic System: Study of the Association Between Serum Measurements and Those Obtained Through Neuroimaging in Healthy Human Adults
Brief Title: Association Between Serum and Neuroimaging Measurements of the GABAergic System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francois Corbin (Other)
Responsible Party: Sponsor-Investigator, Francois Corbin, Full professor, Department of biochemistry, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-5398; 2024-5398 (Other: CÉR CIUSSS Estrie - CHUS)
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: GABAergic System
Keywords: GABAergic system; Neuroimaging; Transcranial Magnetic Stimulation; Magnetic Resonance Spectroscopy
MeSH Terms: interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, single-blind, placebo-controlled design
Who Masked: Participant, Outcomes Assessor
Masking Description: The research team will conduct the randomization and participant code allocation process using REDCap and will dispense the medication or placebo based on the randomization. The placebo will be visibly identical to that of the active medication (i.e. white powder in a gel capsule of the same size and colour as the active medication)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GABA Start Group (Experimental): Participants who are randomly assigned to the GABA start group. These participants receive GABA at the first experimental visit and the placebo at the second experimental visit.
  Interventions: Other: Acute Oral gamma-aminobutyric acid (Natural Health Product in Canada); Other: Acute Placebo
- Placebo Start Group (Experimental): Participants who are randomly assigned to the Placebo start group. These participants will receive a placebo at the first experimental visit and GABA at the second experimental visit.
  Interventions: Other: Acute Oral gamma-aminobutyric acid (Natural Health Product in Canada); Other: Acute Placebo

INTERVENTIONS:
Other: Acute Oral gamma-aminobutyric acid (Natural Health Product in Canada) — 1800 mg (3 capsules of 600mg) of GABA taken at the research center under the supervision of the research team.
  Other Names: GABA
Other: Acute Placebo — A capsule filled with powdered sugar taken under the supervision of the research team.

SUMMARY:
The goal of this study is to better understand the relationship between peripheral and central nervous system measurements of the gamma-aminobutyric acid (GABA) system in otherwise healthy individuals. the main questions it aims to answer are:

1. Does GABA cross the blood-brain barrier?
2. Can peripheral measurements of the GABAergic system be used to study GABA in the brain?

Participants will receive oral GABA and Placebo and undergo blood draws, MRI scans and transcranial magnetic stimulation sessions.

DETAILED DESCRIPTION:
Although gamma-aminobutyric acid (GABA) is the main inhibitory neurotransmitter in the central nervous system in humans, and various pharmacological compounds and natural products aim to modulate it, it is still unknown whether GABA can cross the blood-brain barrier. The present project aims to clarify this issue by comparing measurements obtained in the central nervous system (the brain) with peripheral measurements (serum) following oral administration of the amino acid GABA. This will help determine if peripheral concentrations of GABA in the blood reflect levels in the brain. This would facility studying the GABAergic system in vulnerable clinical populations (such as children or patients with intellectual disabilities) to participate in without resorting to expensive neuroimaging exams and the inclusion of individuals who cannot undergo neuroimaging exams (e.g., claustrophobia, presence of metal in the body). To achieve this, GABA measurements (serum and neuroimaging) will be obtained before and after the oral intake of 1800mg of GABA or a placebo in 30 healthy adults participating in a cross-over, single-blind study with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 35 years old
* Be of right manual dominance
* In good health

Exclusion Criteria:

* Have an implant or pacemaker,
* Having tinnitus,
* Have a history of fainting,
* Have already had an epileptic seizure or have a family history of epilepsy,
* Have a known neurological disease,
* Have a diagnosis of diabetes
* Be under psychotropic medication,
* Have suffered from substance abuse or dependence in the last 6 months,
* Have a neurostimulator,
* Have a splinter or metallic implant in the head or the rest of the body,
* Have a cochlear implant,
* Have an automated injection system implanted (insulin pump),
* Have a transdermal patch,
* Have tattoos in the area to be studied,
* Be pregnant or breastfeeding,
* Being claustrophobic or having other reasons that would prevent the volunteer from tolerating the imaging exam.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Acute GABA consumption on peripheral serum GABA concentrations | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  Serum GABA concentration will be measured before and after acute administration of GABA and placebo.
Impact of Acute GABA consumption on short intracortical inhibition | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  TMS-derived measure of Intracortical inhibition: The degree of decrease of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 70% of resting motor threshold) 2-4 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 millivolt (mV), approximately 120% of resting motor threshold)

SECONDARY OUTCOMES:
Impact of Acute GABA consumption on short intracortical facilitation | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  Transcranial magnetic stimulation (TMS) -derived measure of Intracortical facilitation: The degree of increase of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 80% of resting motor threshold) 12-24 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 mV, approximately 120% of resting motor threshold).
Impact of Acute GABA consumption on GABA concentrations in the brain | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  Estimation of GABA concentrations in the brain from magnetic resonance spectroscopy
Impact of Acute GABA consumption on subjective alertness | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  Subjective alertness will be measured using the Biphasic Alcohol Alertness Scale (BAES). This scale which measures alertness and sedation and is comprised of 6 items, for each item participants rate how they feel from 1 (not at all) to 10 (extremely)
Impact of Acute GABA consumption on objective alertness | Pre-GABA, 40 minutes after acute administration of GABA, Pre-Placebo, 40 minutes after acute administration of Placebo
  Objective alertness will be measured using the psychomotor vigilance task (PVT). This computerised task measures alertness, participants will have to respond to visual cues that are presented at random intervals on the screen.